CLINICAL TRIAL: NCT02831062
Title: Nutritional Therapy to Prevent Progression of Acute Kidney Injury to Chronic Kidney Disease
Acronym: NutriAKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Ravindra Mehta, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151843
Record Dates: First submitted 2016-05-05; First posted 2016-07-13 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease
Keywords: nutrition; progression
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Disease Progression | interventions — Diet, Protein-Restricted; ketosteril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ad lib diet (No Intervention): Patients who have an episode of Stage 2/3 AKI and are followed in a focused post-AKI clinic. Patients will be asked to continue on their regular diet and the protein and caloric ingestion will be recorded at each visit.
- Low Protein Diet + Ketosteril (Experimental): Patients who have an episode of Stage 2/3 AKI and are followed in a focused post-AKI clinic. Patients in this arm will be prescribed a low protein diet (LPD) and +Ketosteril supplementation, containing 0.6 g protein/kg per day, phosphorus 5-10 mg/kg/day, Ketosteril 1 capsule per 5 kg body weight/day divided over three doses (max 8 capsules per dose). Protein and caloric ingestion will be recorded.
  Interventions: Other: low protein diet + ketosteril

INTERVENTIONS:
Other: low protein diet + ketosteril — Patients will follow a diet containing 0.6 g protein/kg per day, phosphorus 5-10 mg/kg/day, Ketosteril 1 capsule per 5 kg body weight/day divided over three doses (max 8 capsules per dose).
  Arms: Low Protein Diet + Ketosteril

SUMMARY:
This study will evaluate patients who have an episode of moderate to severe acute kidney injury (AKI) and are followed in a focused post-AKI clinic. After patients present signs of kidney recovery and before hospital discharge, patients who give consent will be enrolled in the study. At the first post-AKI clinic visit, patients will be randomly allocated to follow a normal (ad-lib) or a low protein diet (LPD) for 3 months. Patients allocated to a LPD will receive a drug called Ketosteril. This drug allows the intake of essential amino acids while minimizing the amino-nitrogen intake, what in excess, can be bad for the recovered kidney. The investigators will evaluate the nutritional parameters and the kidney recovery of all patients and compare these parameters in those two groups.

DETAILED DESCRIPTION:
This is a pilot single center, randomized controlled, trial of patients who have an episode of Stage 2/3 AKI and are followed in a focused post-AKI clinic. Patients will be randomize to either; a. LPD-K diet containing 0.6 g protein/kg per day, phosphorus 5-10 mg/kg/day, Ketosteril 1 capsule per 5 kg body weight/day divided over three doses (max 8 capsules per dose) or b. ad lib diet. Ketosteril should be takes daily during meals and the tablets must not be chewed. Ingestion during meals facilitates proper absorption and the metabolisation into the corresponding amino acids.

After the initial assessment, those randomized to LPD-K will be on this diet for a maximum of 90 days. Additional interventions will include dietary counselling and questionnaire in both groups. We would aim for maintaining serum bicarbonate levels ≥ 22meq/L in both groups.

Evaluation of renal function will be performed using blood and urine tests. In addition, specimens will be collected in a bio-repository, and tested for biomarkers of renal structural damage. Comprehensive nutritional assessment will be performed by a dietitian, along with bioelectrical impedance measurements, blood and urine tests. 24-hour urine urea nitrogen and food records will be used to estimate the protein intake of each individual. Quality of well-being will be assessed using a standardized tool such as Euro Quality of Life (EQ-5D), Charlson Index, and Short Form 8 (SF8) or equivalent. Relevant clinical events (adherence to follow-up, death, hospitalization, renal recovery, repeat AKI episodes) will be tracked throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Duration of stage 2/3 AKI episode ≥ 72 hrs and ≤ 21 days
* Total hospital stay ≤ 21 days

Exclusion Criteria:

* Baseline Chronic Kidney Disease Stage 4 or higher (estimated Glomerular Filtration Rate (eGFR)) <30ml/min/1.73m2) prior to their AKI episode
* Patients dialysis dependent at hospital discharge
* Dialysis dependency > 14 days at time of enrolment
* eGFR exclusion criteria:

  * for patients that required dialysis during hospital stay - measured GFR less than 15ml/min and/or urine output less than 500ml at hospital discharge
  * for patients with known baseline serum creatinine (SCr) - renal recovery with an eGFR more than 80% from baseline at hospital discharge
  * for patients with unknown previous renal function - eGFR > 60ml/min/1.73m2 at time of hospital discharge
* Suspected or biopsy proven glomerulonephritis as cause of AKI
* Obstructive nephropathy as cause of AKI.
* Kidney transplant recipient and patients in the kidney transplant list
* Chronic liver disease
* High likelihood of re-hospitalization or death in the following 6 months, ascertained by physician in charge of the patient.
* Hypercalcemia - Ca > within one standard deviation of reference level upper limit or albumin corrected
* Lactating or pregnant woman or woman planning to become pregnant within the timeframe of the study
* Inability to follow up study procedures for at least 6 months
* Unwillingness to give consent
* Institutionalized individuals (prisoners, significant mental illness, or nursing home residents)
* Body weight <70% or >150% of standard body weight
* History of phenylketonuria or other major disorder of amino acid metabolism
* Hypersensitivity to the active substances or to any of the excipients of Ketosteril.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
feasibility of the LPD-K diet | 6 months
  Feasibility: assess the compliance with diet and drug. Compliance to the assigned protein prescription will be estimated at each visit during the intervention period by nutrient intake data obtained from 3-day food records and the estimated protein intake calculated from urinary nitrogen appearance in 24-hour urine samples. Treatment compliance will be assessed by counting returned tablets.

SECONDARY OUTCOMES:
degree of recovery of renal function | 6 months
  percentage of renal function recovery using baseline estimated GFR as reference. Recovery will be considered as
  * Complete: return of SCr by no less 20% from baseline in patients with known previous renal function. For patients without previous renal function, we will consider complete recovery if measured GFR more or equal to 90ml/min/1.73m2 .
  * Partial: return of SCr less than 20% from baseline in dialysis independent patients. For patients without previous renal function, we will consider partial recovery if measured GFR less than 90ml/min/1.73m2.
rate of recovery of renal function | 6 months
  Slope of renal function recovery using baseline estimated GFR as reference.
safety of the LPD-K diet | 6 months
  Evaluate adverse events related to ketosteril by monitoring serum calcium levels at each visit to determine the development of hypercalcemia Serum calcium levels > 10.5 mg/dl

IPD SHARING:
Plan to Share IPD: No
individual data will not be shared